CLINICAL TRIAL: NCT00988481
Title: Topiramate Augmentation in Bulimia Nervosa Partial Responders
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment.
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Principal Investigator, James Roerig, Principal investigator, Neuropsychiatric Research Institute, Fargo, North Dakota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200909-046
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Bulimia Nervosa
Keywords: Bulimia Nervosa; Topiramate; Augmentation
MeSH Terms: conditions — Bulimia Nervosa | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Topiramate — Topiramate titrated to 200mg/day over four weeks, for ten weeks
  Other Names: Topamax

SUMMARY:
The goal of this study is to generate pilot data exploring the addition of an augmentation (additional) medication to patients suffering from bulimia nervosa who have responded but not had complete symptom resolution with a course of standard medication treatment.

DETAILED DESCRIPTION:
The aim of this study is to determine whether the addition of an augmentation medication (topiramate 200mg/d) will confer additional reductions in symptomatology in BN patients who have received six weeks of standard pharmacological treatment with fluoxetine 60 mg/day or its equivalent and had a partial response but are not in symptomatic remission.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects meeting Diagnostic and Statistical Manual IV edition (DSM-IV) diagnostic criteria for bulimia nervosa (BN).
* Subjects must be between the ages of 18 and 60 years.
* Subjects must currently demonstrate partial response to a standard BN pharmacotherapy treatment.
* Women of child-bearing potential must be practicing an accepted method of birth control (barrier method or oral contraceptive) and have a negative pregnancy test at baseline.
* Subjects must be of good general health by history, laboratory assessment and physical exam.
* Subject's BMI must be >20 and <27 kg/m^2.

Exclusion Criteria:

* Subjects who are allergic to topiramate.
* Subjects who meet DSM-IV criteria for anorexia nervosa.
* Women who are pregnant or nursing at the time of study.
* Subjects experiencing clinically significant, unstable neurological, cardiac, hepatic or renal disease or narrow angle glaucoma.
* Subjects with a history of nephrolithiasis.
* Subjects with a serum potassium <3.0 mmol/L
* Subjects cannot start psychotherapy during the study.
* Subjects currently or with a past history of meeting DSM-IV diagnostic criteria for schizophrenia, schizoaffective disorder, or bipolar disorder.
* Subjects receiving antipsychotic agents, mood stabilizers, antianxiety agents or other non-antidepressant psychotropic agent currently.
* Subjects currently or with a history within the past year of meeting DSM-IV diagnostic criteria for substance abuse.
* Subjects who are experiencing clinically significant suicidal ideation (subjects will be referred to appropriate caregiver).
* Subjects who have participated in an investigational drug study in the past 30 days.
* Subjects who are receiving any prescription medications other than oral contraceptives that will interact with any of the study medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Weekly number of binge eating episodes and purging episodes | Weekly for 10 weeks

SECONDARY OUTCOMES:
Abstinence from BN symptoms | Baseline and endpoint (week 1 and week 10)

CONTACTS AND LOCATIONS:
Overall Officials: James L Roerig, PharmD, BCPP, Principal Investigator — Neuropsychiatric Research Institute, University of North Dakota
Locations (1):
- Neuropsychiatric Research Institute (NRI), Fargo, North Dakota, United States

REFERENCES:
- See also: NRI Official Website — http://www.nrifargo.com/